CLINICAL TRIAL: NCT00287209
Title: Reduction of Atrial Fibrillation Study in Patients Undergoing Coronary Artery Bypass Grafting. (RASCABG 1 Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2003 0245
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2006-02-06 (Estimated); Status verified 2006-02

CONDITIONS: Atrial Fibrillation; Coronary Artery Bypass Grafting
Keywords: RASCABG 1 - study; Postoperative atrial fibrillation; Randomized, controlled trial; Amiodarone
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

INTERVENTIONS:
Drug: Amiodarone

SUMMARY:
The purpose of this study is to determine whether postoperatively oral treatment with high dosis amiodarone for five days after intravenously admitted bolusinfusion will minimize the risk for development of atrial fibrillation after coronary artery bypass grafting.

DETAILED DESCRIPTION:
New-onset atrial fibrillation (AF) after coronary bypass grafting (CABG) is common, with an incidence ranging from 5%-65%.

Although postoperative atrial tachyarrhythmia is often regarded as a temporary problem related to the operation and therefore innocuous, this complication has clinically significant adverse effects on patient outcome.

The purpose of this study was to find a good treatment without severe adverse effects to minimize the incidence of AF and maybe reduced the hemodynamic stress which AF is well known to cause. This would indicate that the risk of developing fatal events like cerebral apoplexy, TCI, AMI and death will be minimized as a result of the improved hemodynamic.

Overall AF is associated with risk of illness and for the development of severe complications as cerebral apoplexy, TCI, AMI and death with a factor 2-3.

There has furthermore been seen a twofold increase in the duration of intensive care unit stay and prolongation of the total hospitalization time with attendant increased hospitalization cost.

The outbreak of AF after CABG has been increasing over the last twenty years. It is speculated that the reason for this rise in incidence is due to the advancing age in the patient populations, more complex cardiac surgery as due to former underestimation of the arrhythmia.

Medical therapy includes various drugs, such as β-blockers, calcium channel blockers, digoxin, sotalol, quinidine, and amiodarone among others, to control heart rate and restore sinus rhythm. Most of these antiarrhythmic agents have significant cardiac and noncardiac adverse effects , why the use of these drugs should be minimized to a short period of time. Amiodarone is well known drug to treat AF and diminish the incidence of AF after CABG operation. So far there has not been any study focusing on postoperative high doses treatment with oral administrated amiodarone. The studies which have been publicized are studies where the drug was administrated intravenously pre-, post- or both pre- and postoperative. Some studies have orally administrated the drug in different regimes11 but no study has yet shown the possible affect of solitarily postoperative administrated high doses amiodarone after an intravenously administrated bolus, with the affect of getting loaded immediately.

ELIGIBILITY:
Inclusion Criteria:

* enlistment for an elective CABG
* age more than 18 years
* willingness to be randomised
* provision of informed consent

Exclusion Criteria:

* enlistment for other types of heart surgery
* earlier heart surgery
* resting heart rate below 40 bpm.
* AV-blockage of any degree
* preoperative atrial fibrillation or flutter
* former known atrial fibrillation or flutter lasting more than one month
* hepatic dysfunction (ALAT > twice the upper normal limit)
* hyperthyroidism
* pregnancy
* breastfeeding
* known adverse reactions to amiodarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2004-01; Study Completion 2005-08

PRIMARY OUTCOMES:
- Time to symptomatic atrial fibrillation, cerebral apoplexy/ transitory cerebral infarction (TCI), acute myocardial infarction (AMI), or death.
- Time to symptomatic or asymptomatic atrial fibrillation, cerebral apoplexy/TCI, AMI or death;
- Time to symptomatic or asymptomatic atrial fibrillation
- Time to symptomatic atrial fibrillation
All measured at postoperative day 7 and 30.

SECONDARY OUTCOMES:
- Length of stay at Skejby Sygehus.
- Length of stay at Skejby Sygehus and local hospital.
- Length of stay at the intensive care unit (ICU) and intermediary unit, Skejby Sygehus

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke E Hjortdal, Professor, Principal Investigator — Department of Cardiothoracic and Vascular Surgery & Institute of Clinical Medicine, Skejby Sygehus, Aarhus University Hospital, DK-8200 Aarhus N, Denmark
Locations (1):
- Department of Cardiothoracic and Vascular Surgery & Institute of Clinical Medicine, Skejby Sygehus, Aarhus University Hospital, Aarhus N, Denmark